CLINICAL TRIAL: NCT00164099
Title: The Role of Synbiotics in Reducing Post-Operative Infections in Patients Undergoing Cardiac Surgery: A Pilot Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Patients would not take product
Sponsor: Beth Israel Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 224-04
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2006-09

CONDITIONS: Surgical Wound Infection; Cystitis; Bacteremia; Pneumonia; Enterocolitis, Pseudomembranous
Keywords: Coronary Artery Bypass; Postoperative Complications; Probiotics; Surgical Wound infection; cystitis; bacteremia; pneumonia; Enterocolitis, Pseudomembranous
MeSH Terms: conditions — Surgical Wound Infection; Cystitis; Bacteremia; Pneumonia; Enterocolitis, Pseudomembranous; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Synbiotic 2000 — See protocol - 4 bacteria, 4 fiber mixture

SUMMARY:
All surgical procedures carry with them the risk of infection. Even a minor infection can extend the hospitalization after cardiac surgery. The average minimum increase in length of stay for a single infection is three days.

One of the many means used to reduce post-operative infections is the preventative, or "prophylactic", administration of antibiotics just before and just after surgery. Because antibiotics, and for that matter surgery itself, alter the body's natural immune and inflammatory responses and the makeup of the bacteria in the intestine, there is a great deal of scientific interest in using the supplementation of bacteria that naturally reside in the intestine. It is felt that by doing so, the alterations in the immune response may be corrected and the patient better able to fight infections. There are studies using probiotics that have demonstrated a reduction in infection rates in patients undergoing abdominal surgery.

Subjects will be patients at high risk for infection including those with any one or more of the following characteristics: over 65 years old, poor heart function (ejection fraction <40), diabetes (insulin dependant or non-insulin dependant), peripheral vascular disease, kidney dysfunction (creatinine level >2mg/dl), obesity (body surface area > 2 m2), low serum protein levels (albumin < 2.5 mg/dl), infection of the heart valve (endocarditis), or on any antibiotics other than standard prophylaxis before surgery.

The safety of these products has been very well established.

Patients who consent to enter the study will receive the synbiotic mix, or a placebo, which comes in a powder that may be mixed with a drink, or washed down into the stomach through the NG tube if the patient is still on a ventilator. Dosing will be initiated within four hours of patient arrival in the Cardiac Surgery Intensive Care Unit and will continue on a twice daily basis for the duration of their admission days. Infection and diarrhea data will be monitored.

DETAILED DESCRIPTION:
Background:

Despite progress in surgical methodology, infections remain one of the most difficult post-operative complications to prevent. In cardiac surgery, the presence of an infection can make the difference between a brief hospital stay and a life-threatening illness. The average minimum increase in length of stay due to a single infection is three days and can extend to months. Nationally, the average rate of deep sternal wound infection is 3% and conduit harvest site infection 1.4%.

Because of the intimate relationship between intestinal bacterial flora and normal gut and immunologic function, current research is investigating the relationship between the preservation or augmentation of certain naturally occurring bacterial strains in the intestine and clinical outcomes, particularly infectious. We propose to examine the efficacy of immediate post-operative supplementation with a product containing four bacterial strains and four different fibers, putatively fuel for bacterial growth, in reducing infections.

Until recently, most studies performed with LAB have selected strains for their palatability and usability in yogurts. For this reason, most studies have been based on LAB, such as Lactobacillus acidophilus, L.casei, L. delbrueckii och Bifidobacillus adolescentis, B.bifidum, B.longum and Bifidobacterium infantis, which are common in yogurts and kefirs. It is only recently that interest has been focused on developing criteria for selecting LAB based on intraluminal biology, such as the ability to adhere to mucus or mucosal cells, the ability to ferment resistant fibers, and antioxidant capacity. For example, L.plantarum, which is often recovered from fermented fruits, vegetables, sourdoughs and silage, has been demonstrated to have a strong ability to adhere to mucosa and to break down resistant fibers. L. plantarum is the commonest LAB in human gastrointestinal tract and has shown the greatest ability of all LAB tested to survive in the gut (106 times that of L.rhamnosus for example) and activate cytokine secretion after passage through the stomach and the small intestine.

The clinical impact of a particular LAB is strongly associated with its ability to colonize the intestinal mucosa. LAB common in dairy products such as yogurts (L.Acidophilus, L.bulgaris and bifidobacteria) have very limited ability to colonize intestinal mucosal cells. L.rhamnosus (GG) and even more so L.plantarum (299) have been shown to remain viable up to 28 days post supplementation. L.plantarum is unique as it uses carbohydrate receptors (mannose) similar to those of gram-negative bacteria (E.coli, Enterobacter, Klebsiella, Salmonella, Shigella, Pseudomonas and Vibrio cholerae). L. plantarum has also been shown to prevent adhesion of enteropathogenic E.coli through induction of mRNA expression for the intestinal mucins MUC2 and MUC3.

Design of the present study 75 consecutive patients deemed at high risk for post-operative infection will be prospectively and blindly randomized to one of the following three groups:

1. Lactic acid bacteria and fermentable fiber
2. Fermentable fiber alone
3. Non-fermentable (placebo)

Sachets containing LAB plus fiber, fiber alone, or placebo will be provided by the manufacturer and will be randomized, coded, and assigned to patients in order. Patients will begin receiving doses within 4 hours of arrival to the CSICU and will remain on treatment twice daily for 14 days.

Data collection Infection control data are collected on all patients undergoing cardiac surgery using established institutional definitions for infections. Incidence of sternal infections, donor site infections, vein harvest site infection, pneumonia, urinary tract infection, catheter and blood stream infections, and clostridium difficile colitis will be considered. In addition, the incidence of diarrhea, defined as stools of liquid or gelatinous consistency, or more than three stools in one day, will be monitored. Data will be collected during hospital stay and at one-month follow-up. Finally, C-reactive protein levels, which are commonly assessed during hospitalizations and used as part of the assessment for coronary risk, will be drawn pre-operatively and four days post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiac surgery, able to consent, and at least one of the following:

  * Age >65 years
  * ejection fraction <=40%
  * diabetes mellitus (insulin requiring and non-insulin requiring)
  * peripheral vascular disease
  * creatinine >=2 mg/dl
  * body surface area >= 2 sq meters
  * endocarditis
  * albumin <=2.5 g/dl
  * on antibiotics for any reason other than operative prophylaxis

Exclusion Criteria:

* Unable to consent
* Not meeting inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Infection | 3 months

SECONDARY OUTCOMES:
Tolerance | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David S Seres, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States